CLINICAL TRIAL: NCT06395038
Title: A Phase I Clinical Trial, Using Interleukin-2 (IL-2) and Abatacept in Patients with Frontotemporal Disorders
Brief Title: IL-2 Plus Abatacept in FTD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Alireza Faridar, Associate Professor, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037661
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-04

CONDITIONS: Frontotemporal Degeneration
MeSH Terms: interventions — Abatacept; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abatacept plus Aldesleukin every 4 weeks (Active Comparator): Subcutaneous abatacept (125 mg) followed by five-day-courses of IL-2 (1MUI/day) every four weeks will be administered for a total of 21 weeks
  Interventions: Drug: Abatacept plus Aldesleukin
- Abatacept plus Aldesleukin every 2 weeks (Active Comparator): Subcutaneous abatacept (125 mg) followed by five-day-courses of IL-2 (1MUI/day) every two weeks will be administered for a total of 21 weeks
  Interventions: Drug: Abatacept plus Aldesleukin

INTERVENTIONS:
Drug: Abatacept plus Aldesleukin — CTLA4IgG plus Low dose Interleukin-2 (Aldesleukin) administration to modify immune responses

SUMMARY:
Neuroinflammation is a significant component of Frontotemporal Disorder (FTD). Our preliminary unpublished data demonstrated that regulatory T cells (Tregs) have a compromised phenotype and reduced suppressive function in FTD patients, skewing the immune system toward a proinflammatory status and potentially contributing to disease progression. Low dose interleukin-2 (IL-2) is now viewed as a very promising immunoregulatory drug with the capacity to selectively expand and restore functional Tregs. Our preclinical data also demonstrated synergistic effect of interleukin-2 and abatacept (CTLA4-IgG) in remodeling immunologic pathways. Abatacept is an FDA approved medication that has been indicated as a monotherapy or concomitantly with other anti-inflammatory drugs to modulate inflammation in autoimmune disorders. This study is a phase I, open-label study to assess safety and tolerability of low dose IL-2 plus abatacept immunotherapy in FTD individuals. In the first part of this study, 5 FTD patients will be recruited. These five individuals will receive subcutaneous abatacept (125 mg) followed by five-day-courses of IL-2 (1MUI/day) every four weeks for a total of 21 weeks (part-1 of the study). If the treatment strategy is safe and well-tolerated, up to 5 additional FTD subjects will be recruited to receive subcutaneous abatacept (125 mg) followed by five-day-courses of IL-2 (1MUI/day) every two weeks for a total of 21 weeks (part 2 of the study).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of probable frontotemporal dementia
2. Male or female age 18 to 86 years
3. If on medications affecting cognition or behaviors (Such as Atypical Antipsychotics, Acetyl Choline Esterase inhibitors), participants must be on stable dosage for at least 4 weeks prior to screening and should remain at a stable dosage during the course of the study. There are no prohibited medications preventing patients from participating in the study.
4. English language speaking
5. Formal education of eight or more years
6. Stable pharmacological treatment of any other chronic conditions for at least 30 days prior to screening
7. A family member or caretaker (study partner) who is expected to be consistently available, administer study drugs of IL-2/abatacept and attend study visits throughout the study. The study partner is also supposed to provide feedback on patient's cognitive and functional status. In the event that the designated study partner is unable to continue participating in the study, the study subject should provide another suitable study partner to ensure the uninterrupted progress of the study.
8. For FTD patients with limited decision-making capacity, the legally authorized representative (LAR) should be present in the decision-making process and trial participation, ensuring they understand the potential risks and benefits, and consent based on the patient's best interest. Extended time for consent will also be considered to ensure comprehension.

Exclusion Criteria:

1. Serious, active bacterial, fungal or viral infection, active or latent tuberculosis
2. History of severe pulmonary dysfunction
3. History of severe cardiac dysfunction defined as left ventricular ejection fraction <40%; a history of non-controlled cardiac arrhythmias; history of cardiac tamponade; Unstable angina or MI in the last 3 months
4. Hypersensitivity or allergy to IL-2 or abatacept
5. History of bowel ischemia/perforation, or GI bleeding requiring surgery
6. Hospitalization or change of chronic concomitant medication within one month prior to screening.
7. History of hemorrhage or infarct or > 3 lacunar infarcts, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, space-occupying lesion (e.g. abscess or brain tumor with the exception of small incidental meningiomas) in prior CT or MRI.
8. Clinical or laboratory findings consistent with:

   1. Other primary degenerative dementia, (dementia with Lewy bodies, Alzheimer's disease, Huntington's disease, Jacob-Creutzfeld Disease, Down's syndrome, Parkinson's disease, etc.)
   2. Seizure disorder
   3. History of infectious, metabolic or systemic diseases affecting the central nervous system (syphilis, Lyme disease, other laboratory values, etc.)
9. Clinically significant, advanced, or unstable disease that may interfere with outcome evaluations, such as:

   1. Respiratory insufficiency
   2. Bradycardia (<45/min.) or tachycardia (>100/min.)
   3. Poorly managed hypertension (systolic >180 mm Hg and/or diastolic >100 mm Hg) or hypotension (systolic <90 mm Hg and/or diastolic <60 mm Hg)
   4. Uncontrolled diabetes defined by HbA1c >8%
   5. Alanine aminotransferase level (ALT) and aspartate aminotransferase (AST) higher than two times normal
   6. Serum creatinine higher than 2 mg/dL
   7. Neutrophil count <1,500/mm3; platelets <100,000/mm3; hematocrit (HCT) <30%.
   8. INR>1.4
10. History of cancer within 3 years of screening with the exception of fully excised non-melanoma skin cancers or non-metastatic prostate cancer that has been stable for at least 6 months.
11. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B
12. Disability that may prevent the patient from completing all study requirements (e.g. blindness, deafness, etc.).
13. Suspected or known allergy to any components of the study treatments.
14. Intake of investigational drug within the previous 30 days or five half-lives of the investigational drug, whichever is longer.
15. Any condition, which in the opinion of the investigator makes the patient unsuitable for inclusion.
16. Contraindication to undergoing an LP including, but not limited to: inability to tolerate an appropriately flexed position for the time necessary to perform an LP; INR >1.4 or other coagulopathy; platelet count of <100,000/μL; infection at the desired lumbar puncture site; taking anti-coagulant medication within 90 days of screening (Note: low dose aspirin is permitted); suspected non-communicating hydrocephalus or intracranial mass; prior history of spinal mass or trauma.
17. Known to be pregnant or lactating, or positive pregnancy test at screening ; This study allows enrolling women of childbearing potential and the treatments may involve unknown risks to the fetus if pregnancy were to occur during the study. This risk is mitigated by requiring proof the participant is not pregnant prior to start of treatment and requiring highly effective contraception during and, for an appropriate interval, after treatment.
18. Lack of reliable study partner.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and the tolerability of abatacept plus IL-2 in FTD patients | 6 months treatment phase
  Number of participants with adverse events and with abnormal laboratory findings (serum chemistry, hematology).

SECONDARY OUTCOMES:
To investigate the impact of low dose IL-2 plus abatacept administration on the blood Treg population in FTD patients | 6 months treatment phase
  Change in Treg percentage out of total # of CD4 cells from baseline to month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes